

NLS Study No.: 665

Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone Sponsor Study No.: ALS-Gd64/001

| STATISTICAL ANALYSIS PLAN | |
|---|---|
| Study Title: | Exploratory evaluation of the potential for long-term retention of Gadolinium (Gd) in the bones of patients who have received Gadolinium based Contrast Agents (GBCAs) according to their medical history. |
| <b>Sponsor Identification:</b> | Navitas Life Sciences GmbH |
| | Hahnstrasse 70 |
| | 60528 Frankfurt, Germany |
| Phase: | Post Authorisation Study / Phase IV |
| Active ingredients of products under evaluation: | Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoteric acid, Gadoversetamide, and Gadoxetic acid |
| Study Number: | ALS-Gd64/001 |
| NLS Study Number: | 665 |
| Responsible Biostatistician: | Sonja Ikemeyer-Fuchs<br>Biostatistician |
| | Navitas Life Sciences GmbH Hahnstraße 70 D-60528 Frankfurt a.M. Tel.: +49-(0)69-66 80 30 0 Fax: +49-(0)69-66 80 30 29 E-mail: Sonja.Ikemeyer-Fuchs@navitaslifesciences.com |
| Date of SAP: | 31JUL2019 |
| Version: | Final 1 |
| Scope: | Final Analysis |



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

### **SIGNATURES**

| Prepared by: | | |
|--------------|------|----------|
| Navitas | Life | Sciences |

GmbH

Author and

Responsible Biostatistician:

Sonja Ikemeyer-Fuchs
Biostatistician

Date:31JUL2019

Review

Dr. Girisha R Medical Writer Date (DD MMM. YYYY)

Sponsor's Representative: Navitas Life Sciences

**GmbH** 

Rajalakshmi S

Manager Biostatistics

Date (DD MMM. YYYY)

Marty Boom

Managing Director

Date (DD MMM. YYYY)

Co-ordinating Investigator:

Professor Christoph Lohmann, MD Universitätsklinikum Magdeburg A. ö. R. Orthopädie - Operatives Zentrum Leipzigerstr. 44 39120 Magdeburg,

Germany

Date (DD MMM. YYYY)



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

#### **SIGNATURES**

| Prepared by: |
|-----------------------|
| Navitas Life Sciences |
| GmhH |

Author and Responsible Biostatistician:

Date:31JUL2019

Review

Medical Writer

Biostatistician

02 AUG 2019 Date (DD MMM, YYYY)

Sponsor's Representative: Navitas Life Sciences GmbH

Rajalakshmi S Manager Biostatistics Date (DD MMM. YYYY)

Marty Boom Managing Director Date (DD MMM, YYYY)

Co-ordinating Investigator:

Professor Christoph Lohmann, MD Universitätsklinikum Magdeburg A. ö. R. Orthopädie - Operatives Zentrum Leipzigerstr. 44 39120 Magdeburg, Germany

Date (DD MMM. YYYY)



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1

Date:31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# **SIGNATURES**

| Prepared by:<br>Navitas Life Sciences<br>GmbH | | |
|---|---|---|
| Author and<br>Responsible Biostatistician: | Sonja Ikemeyer-Fuchs<br>Biostatistician | Date (DD MMM. YYYY) |
| Review | | |
| | Dr. Girisha R<br>Medical Writer | Date (DD MMM, YYYY) |
| Sponsor's Representative:<br>Navitas Life Sciences<br>GmbH | Rajalakshmi S<br>Manager Biostatistics | OR AUG 2019 Date (DD MMM. YYYY) |
| | Marty Boom<br>Managing Director | Date (DD MMM, YYYY) |
| Co-ordinating Investigator: | Professor Christoph Lohmann, MD<br>Universitätsklinikum Magdeburg A. ö.<br>R. Orthopädie - Operatives Zentrum<br>Leipzigerstr. 44 39120 Magdeburg, | Date (DD MMM, YYYY) |

Germany



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1

Date:31JUL2019

Short Title of Study: Long-Term Retention of

Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# **SIGNATURES**

| | 3 | 5 |
|---|---|---|
| Prepared by:<br>Navitas Life Sciences<br>GmbH | | |
| Author and<br>Responsible Biostatistician: | Sonja Ikemeyer-Fuchs<br>Biostatistician | Date (DD MMM. YYYY) |
| Review | Dr. Girisha R<br>Medical Writer | Date (DD MMM. YYYY) |
| Sponsor's Representative:<br>Navitas Life Sciences<br>GmbH | Rajalakshmi S<br>Manager Biostatistics | Date (DD MMM. YYYY) |
| | Marry Boom<br>Managing Director | Date (DD MMM. YYYY) |
| Co-ordinating Investigator: | Professor Christoph Lohmann, MD Universitätsklinikum Magdeburg A. ö. R. Orthopädie - Operatives Zentrum Leipzigerstr. 44 39120 Magdeburg. | Date (DD MMM. YYYY) |

Germany



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1

Date:31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

#### **SIGNATURES**

| Prepared by: | |
|-----------------------|---|
| Navitas Life Science: | 9 |
| GmhH | |

Author and

Responsible Biostatistician:

Biostatistician

Review

Dr. Girisha R Medical Writer Date (DD MMM, YYYY)

Sponsor's Representative: Navitas Life Sciences

GmbH

Rajalakshmi S

Manager Biostatistics

Date (DD MMM, YYYY)

Marty Boom

Managing Director

Date (DD MMM. YYYY)

Co-ordinating Investigator:

Professor Christoph Lohmann, MD Universitätsklinikum Magdeburg A. ö.

R. Orthopädie - Operatives Zentrum

Leipzigerstr. 44 39120 Magdeburg,

Germany

Version No. 3 



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

# Short Title of Study: Long-Term Retention of Gadolinium in Bone Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# 1 TABLE OF CONTENTS

| SIGN | ATURES | 2 |
|---|---|---|
| 1 | TABLE OF CONTENTS 3 | |
| 2 | DOCUMENT HISTORY 5 | |
| 3 | ABBREVIATIONS 6 | |
| 4 | DOCUMENTS | 8 |
| 5 | INTRODUCTION | 8 |
| 6 | | |
| | 6.1 Primary Objectives | 8 |
| | 6.2 Secondary Objectives | 8 |
| 7 | STUDY DESIGN | 8 |
| | <ul><li>7.1 Overview</li><li>7.2 Study Flow-Chart</li></ul> | 8<br>11 |
| | | 12 |
| | 7.3.1 Evaluation Parameters | |
| | 7.3.2 Safety Parameters | 13 |
| 8 | | 13 |
| | 1 | 13 |
| | | 14 |
| | 8.2.1 Group and Stratification Variables | |
| | | 17 |
| | | 17 |
| | 8.5 Data Handling | 17 |
| | 1 | 18 |
| | | 19 |
| | | 19<br>20 |
| | | 20 |
| 9 | | 21 |
| | | 21 |
| | · · | 21 |
| | • | 21 |
| | | 22 |
| | | 22<br>22 |
| | | 22 |
| | | 22 |
| | 9.7 Adverse Events | 23 |
| | 9.8 Other Parameters | 23 |

Version No. 3 



| Sponsor Name: Navitas Life<br>Sciences GmbH | | Short Title of Study: Long-Term Retention of Gadolinium in Bone | |
|---|---|---|---|
| Sta | tistical Analysis Plan (SAP) | | Sponsor Study No.: ALS-Gd64/001 |
| Ver | rsion No.: Final 1 | Date:31JUL2019 | NLS Study No.: 665 |
| 10 | DEVIATION FROM THE STU<br>10.1 Further Deviations | JDY PROTOCOL | 23<br>25 |
| 11 | SOPS FOR ANALYSIS AND | REPORTING | 25 |
| 12 | DATABASE LOCK AND UNI | BLINDING | 26 |
| 13 | REFERENCES | | 26 |
| 14 | LIST OF REPORTED TABLE | S | 26 |
| 15 | LIST OF REPORTED FIGURE | ES | 28 |
| 16 | LIST OF REPORTED SUBJECT | CT DATA LISTINGS | 28 |
| 17 | MOCKUPS OF TABLES AND | SUBJECT DATA LIST | INGS 30 |
| | 17.1 Tables | | 31 |
| | 17.2 Subject Data Listings | | 35 |



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

Short Title of Study: Long-Term Retention of

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

Gadolinium in Bone

# **2** DOCUMENT HISTORY

| Version | Date | Change to previous version |
|---------|-----------|----------------------------|
| Final 1 | 31JUL2019 | No previous version |



Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# **3** ABBREVIATIONS

| ADR | Adverse drug reaction |
|---------|-----------------------------------------------------------|
| AE | Adverse event |
| ATC | Anatomic therapeutic chemical classification |
| BLQ | Below the Limit of Quantification |
| СНМР | Committee for Medicinal Products for Human Use |
| CPS | Counts per Second |
| CSP | Clinical Study Protocol |
| CI | Confidence interval |
| CRF | Case report form |
| CRO | Clinical research organization |
| %CV | Coefficient of Variation (of geometric Mean) % |
| eGFR | Estimated Glomerular Filtration Rate |
| EMA | European Medicines Agency |
| FPFV | First Patient First Visit |
| FAS | Full analysis set |
| Geomean | Geometric Mean |
| Gd | Gadolinium |
| GBCA | Gadolinium based Contrast Agent |
| GLP | Good Laboratory Practices |
| IA | Interim Analysis |
| ICF | Informed Consent Form |
| ICH | International conference on harmonization |
| ICP-AES | Inductively Coupled Plasma - Atomic Emission Spectrometry |
| ICP-MS | Inductively Coupled Plasma - Mass Spectrometry |
| IFC | Informed Consents |
| ITT | Intent-to-treat |
| IP | Investigational product |
| IMP | Investigational medicinal product |
| LLOQ | Lower Limit of Quantification |
| LPLV | Last Patient Last Visit |
| MAH | Marketing Authorization Holder |
| Max | Maximum |
| MedDRA | Medical dictionary for regulatory activities |
| MD | Medicine Doctor |
| Min | Minimum |
| MSc | Master of Science |
| N | Number of non-missing observations |
| Nmiss | Number of missing observations |



Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

| Short Title of Study: Long-Term Retention of |
|----------------------------------------------|
| Gadolinium in Bone |

Sponsor Study No.: ALS-Gd64/001 NLS Study No.: 665

| NSF | Nephrogenic Systemic Fibrosis |
|---|---|
| PPS | Per protocol set |
| PT | Preferred term |
| SAE | Serious adverse event |
| SADR | Serious adverse drug reaction |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SAS | Statistical analysis system |
| SD | Standard deviation |
| SD (geometric) | Geometric standard deviation (re-transformed standard deviation of the logarithms) |
| SOC | System organ class |
| SOP | Standard operating procedure |
| TLF | Tables, Listings and Figures |
| V | Visit |



Short Title of Study: Long-Term Retention of Sponsor Name: Navitas Life Sciences GmbH

Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date:31JUL2019 NLS Study No.: 665

### **DOCUMENTS**

Amended Clinical Study Protocol (CSP) Version 4.0, dated 29 April 2016. Abbreviated Report on the interim analysis, Version 1.0, dated 08 NOV 2018.

### INTRODUCTION

Study ALS-Gd64/001 to evaluate the potential for long-term retention of Gadolinium (Gd) in human bone and skin after administration of Gadolinium based Contrast Agents (GBCAs) and co-factors that may increase the risk of nephrogenic systemic fibrosis (NSF) was requested by the Committee for Medicinal Products for Human Use (CHMP) of the European Medicines Agency (EMA). The study is explorative in nature and will deliver descriptive data on the potential for long-term retention of Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoteric acid, Gadoversetamide, and Gadoxetic acid in human bone and skin.

This Statistical Analysis Plan (SAP) is based on the relevant sections of the amended CSP and includes also the Tables, Listings and Figures (TLF) Specifications. It describes in more detail how the analyses are to be performed and presented.

### STUDY OBJECTIVES

#### 6.1 **Primary Objectives**

To prospectively explore the potential for long-term retention of Gd in bones in subjects who have received a single dose of GBCA or multiple doses of the same GBCA, with moderate or severe renal impairment function or stable normal renal function at the time of GBCA injection.

#### **Secondary Objectives 6.2**

- To evaluate skin samples for concentration of Gadolinium
- To evaluate bone and skin samples for concentrations of calcium, phosphorus, sodium, iron, zinc and potassium
- To evaluate skin samples for any dermatopathological changes that may be associated with NSF
- To describe potential co-factors for NSF, susceptibility factors and drug treatments with potential impact on bone metabolism

#### 7 STUDY DESIGN

#### 7.1 Overview

This is a multicenter, retrospective, prospectively interventional and exploratory, post authorization study, which is conducted globally evaluating the potential for long-term retention of Gd in bones of subjects who received single or multiple doses of GBCAs. The study is retrospective with respect to GBCA administration (no GBCA will be administered to subjects during the study by the investigator), prospective with respect to bone sample collection (taken from surgically removed bone) and both, prospective and interventional regarding skin sample collection. Skin sampling is required for both dermatopathological assessment and quantification of Gd.



NLS Study No.: 665

Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

The study population consists of subjects undergoing an orthopedic procedure, provided that the required amount of trans-operatory collection of bone and skin as defined per-protocol is feasible. All inclusion criteria and no exclusion criteria should be met (please refer to sections 5.1.3, 4.1 and 4.2 of the CSP). Subjects must be aged at least 18 years (or older if required by local regulations) and have received GBCA at least 1 month prior to surgery (test group). Additionally, a group of subjects undergoing hip or knee replacement surgery who have not received GBCA is enrolled (control group).

A minimum of 99 evaluable subjects from centers in America, Europe and Asia have to be enrolled. In the test group at least 84 subjects should be enrolled and in the control group at least 15 subjects should be enrolled. The products assessed should be GBCAs which include one of the active ingredients Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoversetamide or Gadoxetic acid. In the test group at least 13 subjects should be included per GBCA active ingredient group for Gadodiamide, Gadopentetic acid, Gadoversetamide, and Gadoxetic acid and at least 16 subjects should be included per GBCA active ingredient group for Gadobutrol and Gadoteric acid.

Figure 1: Target number of subjects per GBCA



Furthermore, documentation of stable renal function prior to administration of the GBCA is required, and renal function must have been assessed at least once within approximately 3 months prior to GBCA injection. Section 8.2 will describe the stratification plan for all subjects in detail.

The recruitment has started with first subject enrolled in May 2013. Due to difficulties in finding the eligible subjects the recruitment has been extended several times resulting in total recruitment duration of 68 months (from May 2013 until December 2018). End of study for the individual subject is follow-up visit 2 (visit 4) taking place, approximately within 10-14 days after the orthopedic surgery procedure (e.g. hip or knee replacement surgery) at the time of potential stitch removal under normal healing conditions. A detailed schedule of study procedures and assessments is presented in the flow chart of section 7.2.



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date:31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

The study period for each subject includes the scheduled bone and skin sample collection in conjunction with a medically indicated orthopedic surgery procedure. If the subject is scheduled for a second orthopedic surgery procedure (e.g. hip or knee replacement surgery) to be performed within the study period, the subject can continue to participate in the study, provided that the required amount of trans-operatory collection of bone and skin as defined per-protocol is feasible during the second procedure. A second bone and skin sample shall be collected during the second scheduled orthopedic procedure. The overall study period will not be extended in order to obtain the second bone and skin sample collection.

Handling and analysis of trabecular and cortical bone and skin samples will be performed under blinded conditions at central laboratories.



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date: 31JUL2019 Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# **Study Flow-Chart**

Table 7.2.1: Schedule of Procedures and Assessments

| Table 7.2.1: Schedule of Frocedures and A | | | | | | | ~ | | |
|---|---|---|---|---|---|---|---|---|---|
| | Visit 0 | Visit 1 (V1) | <b>Visit 2 (V2)</b> | Visit 3 (V3) | Visit 4 (V4) | If applicable: Subjects receiving a 2 <sup>nd</sup> surgery only | | | |
| | Screening<br>Visit | Baseline<br>(within 3<br>days prior to<br>surgery) | 1 <sup>st</sup> surgery<br>(day 0) | Follow-up 1<br>(3-5 days after<br>surgery) | Follow-up 2<br>(approximately<br>within 10-14 days<br>after surgery) | Visit 5 (V5)* Baseline (within 3 days prior to surgery) | Visit 6 (V6)* 2 <sup>nd</sup> Surgery (within study timeframe) | Visit 7 (V7)* Follow-up 3 (3-5 days after surgery) | Visit 8 (V8)* Follow-up 4 (approximately within 10-14 days after surgery) |
| Subject information and signature on Medical Data Release Form | X | | | | | | | | - |
| Subject information, written informed consent | | Х | | | | | | | |
| Written informed re-consent, if applicable | | | | | | X | | | |
| Demographic data | X | | | | | | | | |
| Diagnosis and medical history | | X | | | | х | | | |
| Inclusion and exclusion criteria | X | X | | | | х | | | |
| Renal status (retrospective with regard to GBCA administrations) | X | | | | | | | | |
| GBCA history / verification of GBCA history | X | Х | Х | | | х | X | | |
| Connection to IWRS for stratified enrolment | | Х | | | | | | | |
| Concomitant diseases and therapies | X | Х | Х | х | х | Х | X | Х | X |
| Study-specific parameters: | | | | | | | | | |
| Bone sample collection | | | Х | | | | X | | |
| Skin sample collection | | | Х | | | | X | | |
| Visual check of wound/scar | | | | X | х | | | X | X |
| Adverse events | | Х | Х | Х | X | Х | X | Х | X |

<sup>\*</sup> Additional visit for subjects scheduled for second orthopaedic surgical procedure within study timeframe In case no second surgery is planned at completion of visit 2, the study ends with the end of the follow-up visit 2 (V4)



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of Sciences GmbH

Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 NLS Study No.: 665 Date: 31JUL2019

#### 7.3 **Parameters**

#### **7.3.1** Evaluation Parameters

#### **Primary Parameter**

- Total Gd concentration in trabecular bone in μg/g
- Total Gd concentration in cortical bone in μg/g

### **Secondary Parameter**

- Total Gd concentration in skin tissue in μg/g
- Gd concentration in bone (trabecular and cortical) and skin as a function of time elapsed between GBCA injection and surgery
- Number of single (one injection of standard dose) or multiple (more than one injection or one injection with higher than standard) doses
- Cumulative dose of GBCA i.e total mmol administered prior to surgery.
- Time elapsed between most recent administration of GBCA [month] and surgery.
- Time of cumulative GBCA doses [months]
- Time intervals of dosing
- eGFR [ml/min/1.73 m<sup>2</sup>]
- Potential co-factors for NSF and susceptibility factors, based on the following data and in the limit of their availability in medical history of the patients:
  - 0 eGFR:
  - cumulative dose of GBCA, 0
  - co-existing vascular, thrombotic and/or pro-inflammatory events
  - serum concentrations of calcium, phosphorus, sodium, iron, potassium and zinc
  - Any event which may have led to Iron mobilization, including concomitant iron drug
  - Cumulative dose of erythropoietin [IU/L]
  - T4 and TSH
- Concomitant drug treatments with potential impact on bone metabolism:
  - biphosphonates
  - estrogens
  - calcitonin 0
  - calcitriol
  - fluoride salts
  - vitamin D
  - corticosteroids
- Concentration of Ca, P, Na, Zn, K and Fe in skin and in tissue of both trabecular and cortical bone, determined by ICP-MS
- Clinical histological evidence of NSF (determined by an experienced dermatopathologist).
- Subjects who have undergone 2 surgeries



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of Sciences GmbH

Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 NLS Study No.: 665 Date: 31JUL2019

#### 7.3.2 **Safety Parameters**

- Adverse event (AE) description
- Onset date/time of AEs
- Resolution date/time of AEs
- Relationship (possibly, probably or certainly related)
  - related to the orthopedic surgery (bone resection included)
  - related to the skin biopsy
  - related to GBCA exposure in the past (e.g. NSF signs after enrolment)
  - related to other health conditions of the subject
- Intensity (mild, moderate, severe)
- Serious (yes, no)

Description of the serious adverse events (SAE)

NSF-like events will be considered medically important events, and thus are serious AEs

- Expectedness (yes, no)
- Outcome of AEs (resolved, resolved with sequelae, not recovered, fatal, unknown)
- Concomitant diseases and medical history
- Previous and concomitant medication

# GENERAL STATISTICAL CONSIDERATIONS

Primary and secondary variables will be analyzed descriptively. No formal hypothesis testing is planned.

#### **Descriptive Statistics** 8.1

The following descriptive statistics will be calculated for continuous data and for ordered categorical data (ordinal data) if applicable:

Summary statistics are displayed with the following digits:

| Description | Characteristic | Number of decimal places |
|---|---|---|
| Count | n | 0 |
| N (number of non-missing measurements) | N | 0 |
| Arithmetic Mean | Mean | As in source + 1 |
| Geometric Mean | GM | As in source + 1 |
| Standard Deviation | SD | As in source + 1 |
| Geometric standard deviation | GSD | As in source + 1 |
| Corresponding %CV | %CV | 2 |
| Minimum | Min | As in source |
| Median | Median | As in source + 1 |
| Maximum | Max | As in source |
| Percentage relative to N | % | 1 * |



Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date: 31JUL2019

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001 NLS Study No.: 665

For ordered categorical data and nominal data, absolute and relative frequencies (in %) will be calculated. A Missing category should be added to any parameter for which information is not available for any subjects and included in all calculations (%).

All relevant medical history conditions and concomitant diseases will be coded in MedDRA and summarized by system organ class and preferred term. The version of the utilized dictionary will be presented as part of the provided tables and listings.

Any disease starting at the date of informed consents or later will be classified as concomitant disease.

All prior and/or concomitant medications and therapies will be coded according to the World Health Organization (WHO) Drug Dictionary according to WHO Preferred Term (ATC level 5). Subjects taking the same medication multiple times will be counted once per medication. The version of the utilized dictionary will be presented as part of the provided tables and listings.

All medication and therapies starting at the date of informed consents (IFC) or later will be classified as concomitant medications and concomitant therapies, whereas, all concomitant medications and therapies starting before the date of IFC will be classified as previous medications and previous therapies. Any previous medications or previous therapies that is still ongoing will be classified as both prior and concomitant medications and prior and concomitant therapies.

All AEs will be presented by primary system organ class and preferred term and sorted alphabetically if not stated otherwise.

All data will be presented in the subject data listings.

If either table or listing does not include any observation, then the following placeholder will be used: "NO DATA CONTRIBUTED TO THIS TABLE / LISTING".

#### 8.2 Grouping and Assignments

Statistical tables will be calculated for all GBCA groups pooled as well as each GBCA group separately and the control group. These will be further stratified according to renal function categories, single/multiple doses (2 groups), and the combination of "renal function with "single / multiple doses".

The CSP did intend to have three different renal function categories:

- Subjects with stable severe renal impairment (eGFR < 30 ml/min/1.73 m<sup>2</sup>)
- Subjects with stable moderate renal impairment (eGFR within the range 30 to 60 ml/min/1.73 m<sup>2</sup>)
- Subjects with stable normal renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>)

<sup>\*</sup> Number of decimal places can be two, if necessary. All table percentages should be rounded to one decimal place if not stated otherwise. If the rounded percentage is 0.0%, then the percentage should be printed as < 0.1%.



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of

Sciences GmbH Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

However, in order to improve recruitment protocol, amendment 3 and finally CSP v.4.0 were established and introduced a change from three renal function groups into two renal function groups. The two subgroups severe renal impairment and moderate renal impairment were combined into "at least moderate impaired renal function" (eGFR <= 60 ml/min/1.73 m<sup>2</sup>) whereas the definition for stable normal renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>) was maintained. As a consequence, recruited subjects showed mostly" moderate" or "normal" impaired renal function, whereas "severe" impaired renal function is very rare. Due to this small sample size (3 subjects in SAF), "severe" and "moderate" impairment will be analyzed as a combined group (at least moderate impaired renal function) in the following. This approach was also followed during the IA and displayed in the IA-CSR.

This study is a multinational, multicenter study. However, due to the small sample size of each stratification group, results will not be further stratified by country or center.

### **8.2.1** Group and Stratification Variables

- GBCA test group or control
- Renal function category (at least moderate impairment (eGFR <= 60 ml/min/1.73 m<sup>2</sup>), stable normal renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>)
- Single (one injection of standard dose) or multiple (more than one injection or one injection with higher than standard) doses of GBCA administered
- Combination of "renal function with "single / multiple doses"
- Elapsed time from first dosing of GBCA until surgery (cumulative dose of GBCA) will be classified and will also be used for stratification.

### 8.2.2 Stratification Plan

#### **GBCA Test Group**

Table 1 and Figure 2 describing targeted number and stratification of subjects for each GBCA group by renal functional status. The numbers reflect the enrolment targets after the introduction of CSP v.4.0. The groups of severe and moderate impaired renal function are combined as explained above **and** in the section 10.

Table 1: Target number of subjects per GBCA and renal function status

| GBCA | Impaired renal function (at least moderate impairment, eGFR $\leq$ 60 ml/min/1.73 m <sup>2</sup> ) | | Stable normal renal function eGFR > 60 ml/min/1.73 m <sup>2</sup> ) | |
|---|---|---|---|---|
| | Single dose | Multiple dose | Single dose | Multiple dose |
| Gadobutrol | 5 | 3 to 5* | 5 | 3 to 5** |
| Gadoteric acid | 5 | 3 to 5* | 5 | 3 to 5** |
| Gadodiamide | 5 | 0 to 5* | 5 | 3 to 5** |
| Gadopentetic acid | 5 | 0 to 5* | 5 | 3 to 5** |
| Gadoversetamide | 5 | 0 to 5* | 5 | 3 to 5** |
| Gadoxetic acid | 5 | 0 to 5* | 5 | 3 to 5** |

<sup>\*</sup> Subjects should be recruited to the Gadodiamide, Gadopentetic acid, Gadoversetamide, and Gadoxetic acid subgroups throughout the study duration up to a maximum of 5, but there is no minimum requirement to reach a specific number of subjects in this subgroup to achieve study completion. At least 3 subjects and a maximum of 5 subjects are required for Gadobutrol and Gadoteric



Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

acid. If the target of 3 subjects is reached, but the study has not yet completed, then recruitment to this subgroup should be continued during the remaining study time.

Figure 2: Stratification of subjects for recruitment purposes by renal functional status and GBCA dosing:



<sup>\*</sup> Depending on the GBCA subgroup

#### **Control Group**

For the control group at least 5 subjects with normal renal function and up to 10 subjects with at least moderate impaired renal function have to be recruited.

<sup>\*\*</sup> At least 3 subjects are required for this subgroup. If the target of 3 subjects is reached, but the study has not yet completed, then recruitment to this subgroup should be continued during the remaining study time, stopping when until 5 subjects have been recruited to this subgroup, or when all other subgroups have reached their minimum target for recruitment, whichever comes first.



Short Title of Study: Long-Term Retention of Sponsor Name: Navitas Life Sciences GmbH

Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

#### 8.3 **Analysis Set**

| Analysis Set | Definition |
|---|---|
| Screening population | All subjects who entered the study |
| Safety analysis set (SAF) | All subjects who have undergone the planned orthopedic surgical procedure |
| Full analysis set (FAS) | All subjects in the SAF for whom Gd measurements from the bone are available |
| Per protocol set (PPS) | All subjects in the FAS who meet the defined requirements of GBCA treatment history, all inclusion and exclusion criteria, and whose tissue samples yield data for Gd in bone (trabecular as well as cortical) and skin. The evaluability of subjects /samples shall be assessed by a blinded |
| | data review prior to final unblinding and analysis. |

#### 8.4 **Protocol Deviation**

The relevant protocol deviations (PD) have to be defined by a systematic data review prior to database closure. For this purpose, PDs that occurred during the study such as deviations of inclusion/exclusion criteria or forbidden concomitant medications will be assessed as 'major' or 'minor' depending on their potential to interfere with the objectives of the study. Listings will be prepared to show the eligibility of all subjects. Comprehensive justification for the classification of a PD as "major" will be given in the integrated clinical study report.

Major protocol deviations and the assessment of analysis sets will be defined during last data review before data base closure. All definitions given in the Minutes of the Final Data Review will be considered in the analysis.

Due to the fact, that the laboratory data for all subjects included in the IA had to be unblinded, these subjects have already been classified before the IA evaluation with regard to PDs.

The list of protocol deviations will be reviewed by the sponsor and finalized before locking the database. The sponsor will identify major protocol violations which will lead to exclusion of subjects from the PPS. Major protocol violations excluded from PPS will be flagged in the protocol violation listing.

#### 8.5 **Data Handling**

There will be no imputation of missing data. All data will be analyzed as they appear in the data base.

Since the geometric mean (the retransformed mean of the logarithmized values) and CV% cannot be calculated in the presence of zero values, the values BLQ were implemented in the IA analysis by half the LLOQ (i.e. 0.025) instead of zero for the calculation of the descriptive statistics. This approach will also be



Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001 NLS Study No.: 665

used for the final analysis. Therefore, values below the limit of quantification (LLOQ) will be replaced by half of the LLOQ (i.e 0.025) instead of zero for the calculation of the descriptive statistics. For adverse events the following rules will be applied:

- AEs with unknown onset date/time will be counted as treatment emergent AEs.
- AEs with unknown end date/time will be counted as an ongoing AE.
- AEs with unknown relationship to GBCA will be counted as related in AE summary tables.
- If for the calculation of a time period the full date format ddmmmyyyy is needed, missing entries will be imputed as follows:
  - o Missing day in start date of a time period is imputed by the first day of the month;
  - o Missing day in stop date of a time period is imputed by the last day of the month;
  - o Missing month in start date of a time period is imputed by January of the year;
  - o Missing month in stop date of a time period is imputed by December of the year;
  - o Missing year is not imputed.

#### 8.6 Sample Size Calculation

Due to the exploratory nature of the study, the sample size was not determined based on formal statistical consideration, but rather on the feasibility of conducting the study as a whole. The study is intended to be analyzed descriptively. No formal hypothesis testing is planned.

There are six groups for active GBCA ingredients (Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoteric acid, Gadoversetamide, and Gadoxetic acid). In each group, two categories of renal function (stable (normal) renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>) versus at least moderate impaired renal (<=60 ml/min/1.73 m<sup>2</sup>) and two subgroups of dosing of GBCA (single / multiple) are to be evaluated.

Per active GBCA ingredient the recruitment targets are defined as follows:

- 5 subjects for stable normal renal function (eGFR > 60 ml/min/1.73 m2) and single dose
- at least 3 subjects and up to 5 subjects for stable normal renal function and multiple doses
- 5 subjects for at least moderate impaired renal function (eGFR <=60 ml/min/1.73 m2) and single dose
- up to 5 subjects for at least moderate impaired renal function (eGFR <=60 ml/min/1.73 m2) and multiple doses. For Gadobutrol and Gadoteric acid, at least 3 subjects are required. For Gadodiamide, Gadopentetic acid, Gadoversetamide, and Gadoxetic acid, there is no requirement to reach a specific number of subjects to achieve study completion.

The total target number of subjects enrolled in these groups will be at least 84.

The number of subgroups in the GBCA-naïve population is two according to renal function category (i.e. at least moderate impairment, and stable normal renal function) and should follow the distribution of the GBCA population. At least five subjects with stable normal renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>) and at least 10 subjects with at least moderate impaired renal function (eGFR  $\leq$  60 ml/min/1.73 m<sup>2</sup>) will



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of

Sciences GmbH Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

be enrolled. Therefore, the total target number of GBCA-naïve subjects enrolled will be at least 15. Consequently, a minimum of 99 subjects in total shall be included in the study.

#### 8.7 Interim Analysis

At the request of the EMA, an interim analysis was to be carried out on all subjects enrolled in the single dose subgroups for Gadobutrol, Gadoteric acid, Gadodiamide, and Gadopentetic acid once at least three subjects had been recruited to the single-dose subgroups for the 4 agents as well as on all subjects of the control group (naïve subjects).

A total of 55 subjects were eligible for the IA. Due to the fact, that the laboratory data for these subjects had to be unblinded, these subjects have already been classified before IA evaluation with regard to PDs. Since one subject had no concentration data available, only 54 subjects were included in the SAF.

To determine the Gd concentration in bone (trabecular and cortical) and skin (expressed as  $\mu g$  Gd / g) the IA based on the SAF and Gd concentrations was descriptively evaluated by:

- Renal function status: stable normal renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>), at least moderate impaired renal function (<=60 ml/min/1.73 m<sup>2</sup>)
- GBCA: Each of the 4 GBCAs (Gadobutrol, Gadoteric acid, Gadodiamide, and Gadopentetic acid) and control

No statistical tests have been calculated.

All data used in the interim analysis have been listed. All listings including subject identifier, GBCA type, renal function, and have been sorted by GBCA type, renal function, and subject identifier. Study investigational sites and analytical laboratories have been blinded to the IA results.

Details on the IA evaluation have been described in the interim SAP and the Abbreviated Interim Analysis Report, Version Final 1.0, dated 20181108.

#### 8.8 Subgroup Analysis

This study was performed as a multinational multicenter study. Due to the small sample size of each stratification group, results will not be further stratified by age or country or center and nor special subgroup analyses will be performed.

The subjects who have undergone two surgeries on study will be analyzed as a subgroup, at least for Gd concentration in bone and skin. Descriptive statistics will be calculated for the difference of Gd concentration in bone (trabecular and cortical) and in skin at the time of first and the time of second surgery. Since the number of subjects in this subgroup is so low, no stratification will be performed.



Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

NLS Study No.: 665

Sponsor Study No.: ALS-Gd64/001

### 8.9 Definitions and Derived Variables

| Definitions and Defived variables | |
|---|---|
| Variable / Term | Definition / Way of calculation |
| Test group | Refers to subjects with GBCA exposure |
| Control | Includes GBCA naïve subjects |
| Stable normal renal function | Stable normal renal function (eGFR > 60 ml/min/1.73 m <sup>2</sup> ), |
| Impaired renal function | Impaired renal function (eGFR <=60 ml/min/1.73 m <sup>2</sup> ) |
| | The groups of sever and moderate impaired renal function are combined as explained in the section 10. |
| Single dose | Only one application of GBCA |
| | (0.1 mmol per kg body weight for Gadobutrol, Gadoteric acid, Gadodiamide, and Gadopentetic acid; 0.025 mmol per kg body weight for Gadoxetic acid) |
| Multiple dose | More than one application of GBCA or one injection with higher than approved standard dose |
| | (0.1 mmol per kg body weight for Gadobutrol, Gadoteric acid, Gadodiamide, and Gadopentetic acid; 0.025 mmol per kg body weight for Gadoxetic acid)) |
| Time between most recent administration of GBCA [month] and surgery | = (Date of surgery – date of most recent GBCA administration +1 day) / 30.25 |
| Time of cumulative GBCA doses [month] | = (Date of surgery – date of first GBCA administration +1 day) / 30.25 |
| Cumulative dose of GBCA (mmol) | = Sum of all administrated GBCA doses |
| Cumulative dose of erythropoietin [IU/L] | = Sum of all administrated erythropoietin doses |

### 8.10 Statistical Software

All statistical analyses will be performed with SAS<sup>®</sup>, Version 9.4 or later. Working instructions are printed in yellow italic text below the shells, e.g.: *Repeat table for PPS* (14.2.2).



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of

Sciences GmbH Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

#### 9 STATISTICAL ANALYSES

The statistical analysis will be carried out for all GBCA groups pooled as well as each GBCA group separately and the control group. They will be further stratified according to renal function category (2 groups), single / multiple doses (2 groups), and the combination of "renal function with "single / multiple doses".

All tables will be programmed for the control group, all GBCA groups pooled as well as for each GBCA group separately. Each table will be presents by all stratification for the renal function categories (2 groups = 2 columns). Repeat tables will be produced by treatment/renal function and dose (single / multiple doses) combined.

Because standard point estimates may be biased when the total number of BLQ values is large (such as when it exceeds 1/3 of the total), the descriptive analysis should only to be calculated if at least 2/3 of the individual data had been measured and found to be above the LLOQ (rationale based on PhUSE\_CSS\_WhitePaper\_PK\_final\_25March2014.pdf).

### 9.1 Subject Disposition

Subject disposition will be tabulated with number and percentages of subjects screened, enrolled, completed according to the protocol, number of surgeries, lost to follow-up or discontinued prematurely. The subjects who prematurely discontinued the study and the reasons for their discontinuation will be presented. Screening failures will be excluded from the analysis but listed in subject data listings.

#### 9.2 Demographic Data and Baseline Characteristics

All Demographic data and baseline characteristics will be displayed for the SAF, FAS and PPS (see definition 8.3).

Demographic data and baseline characteristics will be analyzed using descriptive statistics in summary (mean, SD, median, min and max) or frequency (number and percentage) tables. The following parameters will be analyzed:

- Gender
- Age (years)
- Height (cm)
- Weight (kg)
- Historical use of gadolinium based contrast agent (GBCA)
- Diagnosis of qualifying study indication (affected joint, diagnosis, duration, severity of diagnosis)

#### 9.3 Medical History and Concomitant Diseases

For the SAF medical history conditions and concomitant diseases frequency counts will be summarized by system organ class and preferred term.



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of Sciences GmbH

Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 NLS Study No.: 665 Date: 31JUL2019

#### **Previous and Concomitant Medications**

For the SAF previous and/or concomitant medications and therapies will be summarized in a frequency table, starting at the date of informed consents or later.

#### 9.5 Orthopedic Surgery - Bone and Tissue Sampling

For the SAF number and frequencies will be provided by first and second surgery for:

- Type of surgery (hip replacement surgery, knee replacement surgery shoulder replacement surgery and other orthopedic surgery)
- Surgery site (right, left, other)
- Sample taken (yes, no)
  - o Trabecular bone
  - Cortical bone
  - Skin (for bioanalytics)
  - Skin (for histopathology)

#### 9.6 **Analysis**

#### 9.6.1 **Primary Analysis**

The primary evaluation parameters Gd concentration in bone (trabecular and cortical) will be descriptively tabulated for the control group and each of the 6 GBCAs (Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoteric acid, Gadoversetamide, and Gadoxetic acid) and presented by renal function status: stable normal renal function (eGFR > 60 ml/min/1.73 m<sup>2</sup>) and at least moderate impaired renal function (<=60 ml/min/1.73 m<sup>2</sup>). For mean, SD and %CV the geometric equivalents will be calculated.

The primary analysis will be performed on the full analysis (FAS) and the per protocol set (PPS) (see definitions 8.3).

No statistical tests will be calculated.

#### 9.6.2 **Secondary Analysis**

The secondary evaluation parameter Gd concentration in skin (expressed as µg Gd/g) will be analyzed for the FAS analogously to the primary parameter.

For the following secondary parameter number and percentages or arithmetic summery statistics will be presented for the FAS where applicable.

- Time elapsed between most recent administration of GBCA and surgery in month
- Time of cumulative GBCA doses [month]
- Potential co-factors for NSF and susceptibility factors, based on the following data and in the limit of their availability in medical history of the subjects:
  - eGFR
  - cumulative dose of GBCA
  - co-existing vascular, thrombotic and/or pro-inflammatory events
  - serum concentrations of calcium, phosphorus, sodium, iron, potassium and zinc



Short Title of Study: Long-Term Retention of Sponsor Name: Navitas Life Sciences GmbH

Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

any event which may have led to iron mobilization, including concomitant iron drug

- cumulative dose of erythropoietin
- T4 and TSH.
- Concomitant drug treatments with potential impact on bone metabolism: biphosphonates, estrogens, calcitonin, calcitriol, fluoride salts, vitamin D, corticosteroids.
- Concentration of Ca, P, Na, Zn, K and Fe in skin and in tissue of both trabecular and cortical bone determined by ICP-MS.

No statistical tests will be calculated.

#### 9.7 **Adverse Events**

Safety analysis will be performed for the SAF and will be included the investigation of adverse events (AEs), serious adverse events (SAEs) and adverse drug reactions (ADRs) as well as serious adverse drug reactions (SADR)s.

For all AEs occurring after enrolment, a summary containing the following counts and percentages of subjects will be presented by treatment:

- Number of AEs
- Number and percentage of subjects with at least one AE
- Number and percentage of subjects with at least one AE:
  - related to the orthopedic surgery (bone resection included)
  - related to the skin biopsy
  - related to GBCA exposure in the past (e.g. NSF signs after enrolment)
  - related to other health conditions of the subject
- Number and percentage of subjects with expectedness for potential AEs in response to GBCA exposure in the past (e.g. NSF signs after enrolment)
- Number and percentage of subjects with AEs by intensity
- Number and percentage of subjects with SAEs
- Number and percentage of subjects who died
- Number and percentage of subjects who discontinued due to AE

Further, all AEs, SAEs, ADRs and SADRs will be summarized in a frequency table by MedDRA system organ class and preferred term. The version of the utilized dictionary will be presented as part of the provided tables and listings.

#### 9.8 **Other Parameters**

Not applicable.

### 10 DEVIATION FROM THE STUDY PROTOCOL

The planned analysis will be performed according to the study protocol, its amendments and this statistical analysis plan. If there are contradictions between the study protocol or its amendments and this statistical



Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001 NLS Study No.: 665

analysis plan, the analysis will be performed according to this analysis plan. Any deviation from the planned analysis according to the study protocol has to be described in the integrated report.

The differences between study protocol and statistical analysis plan are summarized in the following table:

| Change | Study protocol | Statistical analysis plan |
|---|---|---|
| | | Will be changed to: |
| Wording in CSP | GdCA | GBCA |
| | Impaired renal function (eGFR <30 ml/min/1.73 m² (severe) and ≥30 to <=60 ml/min/1.73 m² (moderate)) | At least moderate impaired renal function (eGFR <=60 ml/min/1.73 m²) In order to improve recruitment CSP amendment 3 introduced a change from three renal function groups into two renal function groups. The two subgroups severe renal impairment and moderate renal impairment were combined into "at least moderate impaired renal function" (eGFR <= 60 ml/min/1.73 m²) whereas the definition for stable normal renal function (eGFR > 60 ml/min/1.73 m²) was maintained. As a consequence, recruited subjects showed mostly" moderate" or "normal" impaired renal function, whereas "severe" impaired renal function is very rare. Due to small sample size (3 patients in SAF), "severe" and "moderate" impairment.needs to be combined |
| Wording in CSP used in section 8.1.2 | Statistical tables will compare<br>all GdCA groups pooled as<br>well as each GdCA group<br>separately versus the control<br>group. | Statistical tables will be calculated for all GBCA groups pooled as well as each GBCA group separately and the control group. |



Sciences GmbH

Statistical Analysis Plan (SAP)


| LIFE SCIENCES |
|-----------------------------------------------------------------|
| Short Title of Study: Long-Term Retention of Gadolinium in Bone |

NLS Study No.: 665

Sponsor Study No.: ALS-Gd64/001

| Change Study protocol | | Statistical analysis plan Will be changed to: |
|---|---|---|
| | They will be further stratified according to renal function category (3 groups), single / multiple doses of all subjects (2 groups), and the combination of "renal function with "single / multiple doses". | They will be further stratified according to renal function category (2 groups), single / multiple doses of all subjects (2 groups), and the combination of "renal function with "single / multiple doses". |
| | The number of subgroups in the GdCA-naïve population is 3 according to renal function category (i.e. severe or moderate impairment, and stable normal renal function). | The number of subgroups in the GdCA-naïve population is 2 according to renal function category (at least moderate impairment, and stable normal renal function). |

#### 10.1 Further Deviations

In the IA report as compared to the IA SAP is the replacement of values BLQ defined by half of the LLOQ (i.e 0.025) instead of zero for the calculation of the descriptive statistics because in the presence of zero values, the geometric mean (the re-transformed mean of the logarithmized values) and %CV cannot be calculated. This procedure will also apply here (see Section 8.5)

### 11 SOPS FOR ANALYSIS AND REPORTING

Navitas Life Sciences standard operating procedures are to be used for this analysis.

The following SOPs are to be used

| Title |
|---|
| ICH Topic E9(CPMP/ICH/363/96) "Note for Guidance on Statistical Principles for Clinical Trials" |
| NLS.STAT.ALL.SOP.005 – Preparation of SAP |
| NLS.STAT.ALL.SOP.007 - Create raw datasets, derived datasets and archive data |
| NLS.STAT.ALL.SOP.009 – Perform Statistical Analysis and Generate Tables, Graphs and Listings |
| NLS.STAT.ALL.SOP.011 – Validating SAS programs |

The structure of post-text-tables and the appendices will be in accordance with the ICH guideline E3.



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of

Sciences GmbH Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

### 12 DATABASE LOCK AND UNBLINDING

The SAP will be finalized prior to database lock or any unblinding of study team members. After the data cleaning process is finalized according to the data management plan (DMP) and the assignment of subjects to the analysis sets is agreed and signed by the sponsor, the study data base will be locked. SAS datasets will be extracted from the study data base as described in the DMP.

### 13 REFERENCES

European Medicines Agency (EMA). Guideline on bioanalytical method validation (2011). http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientificguideline/2011/08/WC500109686.pd f. Accessed 24 Oct 2018. Further references are given in the study protocol.

### 14 LIST OF REPORTED TABLES

Tables will be numbered within their section in ascending order. In this SAP the numbering of all TLFs is done according to the ICH guidelines.

Note that TLFs in this SAP may differ slightly from the layout of the IA SAP tables. That is due to the fact that the IA SAP was created according to the old ECRON ACUNOVA standard and the current SAP is written according to the Navitas Life Science standard.

| No. | Title | Analysis Set | Corresponding |
|---|---|---|---|
| | | | Table in the IA |
| 14.1 | <b>Subject Disposition</b> | All Subjects | |
| 14.1.1 | Subject Disposition | Applicable | A 1 |
| 14.2 | Demographic Data and Baseline<br>Characteristics | SAF, FAS,<br>PPS | |
| 14.2.1 | Demographic Characteristics | Applicable | A 2.1 – A 2.5 |
| 14.2.2 | Baseline Characteristics - Diagnosis of<br>Qualifying Study Indication | Applicable | Not Applicable |
| 14.3 | Medical History and Concomitant<br>Diseases | SAF | |
| 14.3.1 | Relevant Medical History | Applicable | Not Applicable |
| 14.3.2 | Concomitant Diseases | Applicable | Not Applicable |
| 14.4 | Previous and Concomitant<br>Medications | SAF | |
| 14.4.1 | Prior Medication and Therapies | Applicable | Not Applicable |
| 14.4.2 | Concomitant Medication and Therapies | Applicable | Not Applicable |
| 14.5 | Orthopedic surgery | SAF | |



Sciences GmbH

Statistical Analysis Plan (SAP)


| Short Title of Study: Long-Ter | m Retention of |
|--------------------------------|----------------|
| Gado | linium in Bone |

Sponsor Study No.: ALS-Gd64/001 NLS Study No.: 665

No. Title **Analysis Set** Corresponding Table in the IA 14.5.1 Bone and Tissue Sampling **Applicable** Not Applicable FAS, PPS 14.6 **Analysis** 14.6.1 **Primary Analysis Applicable** 14.6.1.1 Gadolinium Concentration in Trabecular **Applicable** A 3.1.1 – A 3.1.5 Bone by Renal Function Status A 3.1.7 – A 3.1.11 14.6.1.2 Gadolinium concentration in Cortical Applicable Bone by Renal Function Status PPS 14.6.2 **Secondary Analysis** 14.6.2.1 Gadolinium concentration in Skin by **Applicable** A 3.2.1 – A3.2.5 Renal Function Status 14.6.2.2 Time between last Administration of Applicable Not Applicable GBCA and the Date of Tissue Sample Collection 14.6.2.4 Individual eGFR values Not Applicable **Applicable** Potential Co-Factors for NSF and 14.6.2.5 Applicable Not Applicable Susceptibility Factors Concomitant Drug Treatments with 14.6.2.6 Applicable Not Applicable Potential Impact on Bone Metabolism 14.6.2.7 Concentration of Ca, P, Na, Zn, K and Fe Not Applicable Applicable in skin and in tissue of both trabecular and cortical bone determined by ICP-MS Histopathological evaluation of skin 14.6.2.8 **Applicable** Not Applicable samples (taken at time of surgery / surgeries) with regard to the possibility of findings associated with NSF 14.7 **Adverse Events** SAF, FAS, **PPS** 14.7.1 Summary of Adverse Events Not Applicable Applicable 14.7.2 Adverse Events by System Organ Class Not Applicable Applicable and Preferred Term (MedDRA Version 14.7.3 GBCA Related Adverse Event by System Applicable Not Applicable Organ Class and Preferred Term (MedDRA Version x.x) 14.7.4 Serious Adverse Events by System Applicable Not Applicable Organ Class and Preferred Term (MedDRA Version x.x)



Sponsor Name: Navitas Life Short Title of Study: Long-Term Retention of

Sciences GmbH Gadolinium in Bone

Statistical Analysis Plan (SAP) Sponsor Study No.: ALS-Gd64/001

Version No.: Final 1 Date: 31JUL2019 NLS Study No.: 665

| No. | Title | Analysis Set | Corresponding |
|---|---|---|---|
| | | | Table in the IA |
| 14.7.5 | GBCA Related Serious Adverse Events<br>by System Organ Class and Preferred<br>Term (MedDRA Version x.x) | Applicable | Not Applicable |
| 14.7.6 | Serious Adverse Events and Death by<br>Subject (MedDRA Version x.x) | Applicable | Not Applicable |

## 15 LIST OF REPORTED FIGURES

Not applicable.

# 16 LIST OF REPORTED SUBJECT DATA LISTINGS

In general, subject data listings should include all subjects with data. The numbering of all TLFs is following the ICH guidelines.

To display all necessary subject data for the IA there was only one subject data listing created. Since this SAP will display all available data for all included subjects, there will be no equivalent listing to the IA SAP. The provided IA listing is a combination out of subject data listing 16.2.2.1, 16.2.6.1 and 16.2.6.2.

| No. | Title |
|---|---|
| 16.2.1 | Subject Disposition |
| 16.2.1.1 | Subject Enrolled but Surgery did not take place |
| 16.2.1.2 | Subjects who Discontinued Prematurely |
| 16.2.1.3 | Subjects Applying for Interim Analysis |
| 16.2.1.4 | Protocol Violations |
| Preface A | List of Inclusion and Exclusion Criteria |
| 16.2.1.5 | Eligibility Criteria |
| 16.2.2 | Demographic Data and Baseline Characteristics |
| 16.2.2.1 | Demographic Characteristics |
| 16.2.2.2 | Baseline Characteristics - Diagnosis of Qualifying Study Indication |
| 16.2.3 | Medical History and Concomitant Diseases |
| 16.2.3.1 | Relevant Medical History and Concomitant Disease(S) |
| 16.2.4 | Previous and Concomitant Medication |
| 16.2.4.1 | Prior and/or Concomitant Medication and Therapy |
| 16.2.5 | Orthopedic surgery |



Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1

Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

Date: 31JUL2019 NLS Study No.: 665

| No. | Title |
|---|---|
| 16.2.5.1 | Bone and tissue sampling by Surgery Number |
| 16.2.6 | Analysis |
| 16.2.6.1 | Gadolinium Contrast Agent (GBCA) |
| 16.2.6.2 | Dosing Timepoints and Intervals |
| 16.2.6.3 | Vascular, Thrombotic and/or Proinflammatory Events |
| 16.2.6.4 | Concomitant Drug Treatments with Potential Impact on Bone Metabolism |
| 16.2.6.5 | Serum Concentrations |
| 16.2.6.6 | Iron Mobilization Events |
| 16.2.6.7 | Disorders Related to T4/Tsh |
| 16.2.6.5 | Erythropoietin Treatments |
| 16.2.6.6 | Histopathological evaluation of skin samples |
| 16.2.7 | Adverse Events |
| Preface B | Legends to Adverse Events |
| 16.2.7.1 | Adverse Events |
| 16.2.7.2 | Original Onset and End Dates and Times of Adverse Events |
| 16.2.8 | General Checks |
| 16.2.8 | General Checks by Visit |
| 16.2.9 | End of Study |
| 16.2.9 | End of Study |



Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

### 17 MOCKUPS OF TABLES AND SUBJECT DATA LISTINGS

Please note: Yellow resp. cursive texts are working advices.

#### In General:

• Required margins: at least 1.0 cm on the upper and lower margin and at least 1.5 cm on the left and right sides. All tables and listings will be landscape and centered format. All figures will be landscape and centered format, unless portrait orientation suggests that the information presented is easier to interpret.

All output should have the following header at the upper left margin:

<Sponsor>

Protocol No.: <Protocol No.>

and the following header at the upper right margin:

<Draft/Final Version>, ddmmmyyyy

Page n of N

- Tables/appendices/listings should be internally paginated (i.e., page numbers should appear sequentially within each table). The name of the SAS program used to generate the output shall be displayed in the lower left corner. SAS Monospace, font size 8 will be used, although the mockup below would indicate differently.
- Tables of Contents will be generated separately for Tables and Listings, listing numbers and titles. A file separate from Tables and Listings output must be produced. TOC pages will bear the standard header.

#### Tables in general:

- Each table will present all types of renal function in separate columns and next to each other. If necessary, add a column for total.
- If applicable tables will be repeated by treatment (Control, GBCA-Overall, Gadobutrol, Gadodiamide, Gadopentetic acid, Gadoteric acid, Gadoversetamide, and Gadoxetic acid) and by treatment and dose (single/multiple) separately.

#### Data Listings in general:

• All Listings should be - paged by treatment and sorted by renal function, subject and actual date and time.

Use the appropriate table type as shown below. For more detail description refer to NLS Catalog for Mock ups to support the SAP.

Version No. 3 



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

### 17.1 Tables

Navitas Life Sciences GmbH

Protocol No.: ALS-Gd64/001 Version 4.0

Date: ddmmmyyyy

Page n of N

Table of Contents

| Table Number | Title | Analysis Set |
|--------------|---------------------|--------------|
| Table 14.1 | Subject Disposition | All Subjects |

Please, provide as separate file

YYYYY.sas SAS Version: XX

Version No. 3 



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# **Type 1: Frequencies**

Navitas Life Sciences GmbH

Protocol No.: ALS-Gd64/001 Version 4.0

Date: ddmmmyyyy Page n of N

Table 14.x.x Title

Analysis Set: SAF, FAS, PPS, Treatment T Single Dose

| Characteristic | Total<br>(N=xxx) | Stable Normal Renal Function<br>(eGFR > 60 ml/min/1.73 m2)<br>(N=xxx) | At least Moderate Impaired Renal Function<br>(eGFR <= 60 ml/min/1.73 m2)<br>(N=xxx) | Missing Renal<br>Function |
|---|---|---|---|---|
| Variable 1 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Sub-Category 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) | XX (XX.X) |
| Sub-Category 2 | | ••• | ••• | |
| Sub-Category 3 | | ••• | ••• | |
| | | ••• | ••• | |
| Category 2 | | ••• | ••• | |
| Sub-Category 4 | | ••• | ••• | |
| Sub-Category 5 | | | ••• | |
| | | | ••• | |
| Variable 2 n (%) | | ••• | ••• | |
| Category 1 | | ••• | ••• | |
| Sub-Category 1 | | ••• | ••• | |
| | | | ••• | |

Footnotes

Use Treatment, Dose Category and Sub-Category only if necessary. For each population start a new page. If necessary, add footnotes.

YYYYY.sas SAS Version: XX

Version No. 3 



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

### **Type 2: Summary Statistics**

Navitas Life Sciences GmbH

Protocol No.: ALS-Gd64/001 Version 4.0

Date: ddmmmyyyy Page n of N

Table 14.x.x Title

Analysis Set: SAF, FAS, PPS Treatment - Single Dose

At least Moderate Impaired Renal Function Stable Normal Renal Function Missing Renal Characteristic (eGFR > 60 ml/min/1.73 m2) $(eGFR \le 60 \text{ ml/min}/1.73 \text{ m2})$ Total Function Variable 1 Category 1 Sub-Category 1 XX XX XX XX Mean xx.xxx.xXX.XXX.X . . .

Sub-Category 2

. . .

Variable 2 Category 1

n

Footnotes

Use Treatment, Dose, Category and Sub-Category only if necessary. Provide all statistics according to 8.1. For each population start a new page. If necessary, add footnotes.

YYYYY.sas SAS Version: XX

Version No. 3 



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

# Type 3: Frequencies and Summary Statistics Combined

Navitas Life Sciences GmbH

Protocol No.: ALS-Gd64/001 Version 4.0

Date: ddmmmyyyy Page n of N

At least Moderate Impaired Renal

Table 14.x.x Title

Stable Normal Renal

Analysis Set: SAF, FAS, PPS Treatment

| Characteristic | Total | Function (eGFR > 60 ml/min/1.73 m2) | Function (eGFR <= 60 ml/min/1.73 m2) | Missing Renal<br>Function |
|---|---|---|---|---|
| Variable 1 n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Category 1 | | ••• | ••• | |
| Sub-Category 1 | | | ••• | |
| Sub-Category 2 | | | ••• | |
| Sub-Category 3 | | ••• | | |
| Category 2 | | ••• | | |
| Sub-Category 4 | | | ••• | |
| Sub-Category 5 | | ••• | ••• | |
| Variable 2 | | | | |
| Category 3 | | | | |
| Sub-Category 1 | | | | |
| n | | | ••• | |
| Mean | | | ••• | |
| SD | | | ••• | |

Footnotes

Use Treatment, Category and Sub-Category only if necessary. Provide all statistics according to 8.1. For each population start a new page. If necessary, add footnotes.

YYYYY.sas SAS Version: XX



Sciences GmbH

Statistical Analysis Plan (SAP)

Version No.: Final 1 Date: 31JUL2019 Short Title of Study: Long-Term Retention of Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

### 17.2 Subject Data Listings

All variables out of all available case report forms (CRFs) will be listed. Each subject data listing will be paged by treatment and renal function will be the first column followed by Subject ID. The Subject Data Listing which is presented below after table of contents is only an example, it will be expended according to study objectives and CRF.

Date: ddmmmyyyy Navitas Life Sciences GmbH Page n of N

Protocol No.: ALS-Gd64/001 Version 4.0

Table of Contents

| Listing Number | Title |
|----------------|-------|
| 16.2.1.1 | ••• |
| • • • | ••• |

Please, provide as separate file.

YYYYY.sas SAS Version: XX

Version No. 3 



Sponsor Name: Navitas Life

Sciences GmbH

Statistical Analysis Plan (SAP)


Short Title of Study: Long-Term Retention of

Gadolinium in Bone

Sponsor Study No.: ALS-Gd64/001

NLS Study No.: 665

Navitas Life Sciences GmbH

Protocol No.: ALS-Gd64/001 Version 4.0

Date: ddmmmyyyy Page n of N

Subject Data Listing 16.2.x.x
Title

| | | | | 110 | LC | | | |
|---|---|---|---|---|---|---|---|---|
| Treatment. | <mark>: xxxxx</mark> | | | | | | | |
| Renal | Subject | | | | | | | |
| Function | ID | | <br> | | | <br> | <br> | <br> |
| xxxx | xxxx | | <br> | | | <br> | <br> | <br> |
| | xxxx | | <br> | | | <br> | <br> | <br> |
| xxxxxx | xxxx | | <br> | | | <br> | <br> | <br> |
| | xxxx | | <br> | | | <br> | <br> | <br> |
| | | • • • | <br> | | | <br>• • • | <br>• • • | <br> |

YYYYY.sas SAS Version: XX